CLINICAL TRIAL: NCT04591886
Title: Randomized Controlled Trial of the Peer-Delivered "Mind. Body. Voice." Eating Disorder Prevention Program Among High School Women
Brief Title: The Peer-Delivered "Mind. Body. Voice." Program for High School Women
Acronym: mbv
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, Sona Dimidjian, PI, University of Colorado, Boulder
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18-0007-02
Record Dates: First submitted 2020-10-10; First posted 2020-10-19 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Eating Disorders in Adolescence
Keywords: Eating disorder prevention; Female; Adolescence; Peer delivery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mind. body. voice. (Experimental): The 10-week mind. body. voice. program
  Interventions: Behavioral: mind. body. voice.
- Control (No Intervention): Assessment-only control

INTERVENTIONS:
Behavioral: mind. body. voice. — The mbv program consists of 10 weekly sessions that include a variety of practices, including: cognitive dissonance exercises, contemplative practices, guided discussion and community building.
  Arms: mind. body. voice.

SUMMARY:
This study will evaluate the impact of a program (called mind. body. voice. or "mbv") that was collaboratively designed by youth, educators, and researchers, informed by the Body Project (Becker et al., 2013; Stice et al., 2019), Youth Participatory Action Research, and an extended co-design process. The study evaluates the impact of the mbv program on key aspects of mental health and well-being; specifically, body image and disordered eating symptoms, identity and agency, social and self-constructs, physical health and mood at five time points over the course of a year. Students will be recruited from two high schools and will be randomized to receive the mbv program or an assessment-only control group.

DETAILED DESCRIPTION:
Eating disorders have the highest mortality rate of any psychiatric condition and are the second leading cause of mental health disability among young women. Given that eating disorders have their peak onset during adolescence (ages 16-19), prevention efforts among adolescent women are critical in order to avert the onset of these chronic and disabling disorders. The mbv program targets body image and appearance related pressures, awareness of body sensations, and agency and community building skills.The program consists of 10 weekly sessions and is delivered by peer facilitators. This study will implement and evaluate the mbv program at the high school level in order to examine the extent to which the program influences young women's mental health and well-being, particularly related to eating disorder risk factors and symptoms.

Utilizing a longitudinal randomized controlled trial, the study seeks to address the following aims:

1. To examine the impact of the mbv program on key aspects of mental health and well-being; specifically, body image and disordered eating symptoms, identity and agency, social and self- constructs, physical health and mood among participating high school women.
2. To explore young women's experiences of participating in the program, including strengths and limitations and perspectives on specific activities.

ELIGIBILITY:
Inclusion Criteria:

* High school women, grades 9-12

Exclusion Criteria:

* Prior participation in the Body Project

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — identify as female
Enrollment: 120 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Dieting Behavior and Restraint | baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline), 6-month post intervention follow-up, 1-year post intervention follow-up
  Self-report measure of dieting behavior and restricted eating (scale 1-5 with higher scores indicating higher levels of dieting and restriction)
Change in Body Dissatisfaction Scale | baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline), 6-month post intervention follow-up, 1-year post intervention follow-up
  Self-report measure of body dissatisfaction (scale 1-5 with higher scores indicating higher levels of dissatisfaction)
Change in Objectified Body Consciousness Scale | baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline), 6-month post intervention follow-up, 1-year post intervention follow-up
  Self-report measure of body monitoring and surveillance (scale 1-5 with higher scores indicating higher levels of body surveillance)
Change in Ideal Body Stereotype Scale | baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline), 6-month post intervention follow-up, 1-year post intervention follow-up
  Self-report measure of internalization of ideal body stereotypes (scale 1-5 with higher scores indicating higher levels of internalization)
Change in Body Appreciation Scale | baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline), 6-month post intervention follow-up, 1-year post intervention follow-up
  Self-report measure of body appreciation (scale 1-5 with higher scores indicating higher levels of appreciation)
Change in Social Contribution Scale | baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline), 6-month post intervention follow-up, 1-year post intervention follow-up
  Self-report measure of sense of contributing to society (scale 1-5 with higher scores indicating higher levels of contribution)
Change in Engaged Living Scale | baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline), 6-month post intervention follow-up, 1-year post intervention follow-up
  Self-report measure of values-based living (scale 1-5 with higher scores indicating higher levels of living based on values)
Change in Multidimensional Assessment of Interoceptive Awareness | baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline), 6-month post intervention follow-up, 1-year post intervention follow-up
  Self-report measure of somatic awareness (scale 1-5 with higher scores indicating higher levels of somatic awareness)
Change in Self-Liking and Self-Competence Scale | baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline), 6-month post intervention follow-up, 1-year post intervention follow-up
  Self-report measure of how much one likes oneself and considers oneself competent (scale 1-5 with higher scores indicating higher levels of self-liking and self-competence)
Change in Proactive Coping Scale | baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline), 6-month post intervention follow-up, 1-year post intervention follow-up
  Self-report measure of ability to succeed (scale 1-5 with higher scores indicating higher levels of proactive coping)
Change in Self-Efficacy Scale | baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline), 6-month post intervention follow-up, 1-year post intervention follow-up
  Self-report measure of effectiveness in handling challenges and achieving goals (scale 1-5 with higher scores indicating higher levels of self-efficacy)
Change in Internalization of Media Appearance Ideals | baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline), 6-month post intervention follow-up, 1-year post intervention follow-up
  Self-report measure of internalized appearance ideals in the media (scale 1-5 with higher scores indicating higher levels of internalization)
Change in Sociocultural Pressures Around Appearance | baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline), 6-month post intervention follow-up, 1-year post intervention follow-up
  Self-report measure of sociocultural pressures related to appearance (scale 1-5 with higher scores indicating higher levels of pressure)
Change in Peer Influence on Appearance Concerns | baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline), 6-month post intervention follow-up, 1-year post intervention follow-up
  Self-report measure of influence of peers on appearance concerns (scale 1-5 with higher scores indicating higher levels of peer influence)
Change in Group Belonging Scale (intervention group only) | baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline), 6-month post intervention follow-up, 1-year post intervention follow-up
  Self-report measure of sense of anticipated (baseline) and experienced (follow-up) belonging with intervention program group (scale 1-7 with higher scores indicating higher levels of belonging)
Change in Self-Compassion Scale | baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline), 6-month post intervention follow-up, 1-year post intervention follow-up
  Self-report measure of compassion for oneself (scale 1-5 with higher scores indicating higher levels of self-compassion)
Change in Belonging Scale | baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline), 6-month post intervention follow-up, 1-year post intervention follow-up
  Self-report measure of general sense of belonging (scale 1-5 with higher scores indicating higher levels of belonging)

SECONDARY OUTCOMES:
Change in Eating Disorder Symptoms and Diagnoses | baseline, post-intervention (10 weeks after baseline),
  Interview data on eating disorder symptoms and diagnoses (Kiddie Schedule for Affective Disorders and Schizophrenia, Eating Disorder Supplement)
Change in Eating Attitudes Test 26 | baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline), 6-month post intervention follow-up, 1-year post intervention follow-up
  Self-report measure of disordered eating behaviors (scale 1-6 with higher scores indicating higher levels of disordered eating)
Change in Generalized Anxiety Disorder 7 | baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline), 6-month post intervention follow-up, 1-year post intervention follow-up
  Self-report measure of anxiety (scale 1-4 with higher scores indicating higher levels of anxiety)
Change in Patient Health Questionnaire 9 | baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline), 6-month post intervention follow-up, 1-year post intervention follow-up
  Self-report measure of depression (scale 1-4 with higher scores indicating higher levels of depression)
Change in UCLA Loneliness Scale | baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline), 6-month post intervention follow-up, 1-year post intervention follow-up
  Self-report measure of loneliness (scale 1-4 with higher scores indicating higher levels of loneliness)
Change in Positive and Negative Affect Scale | baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline), 6-month post intervention follow-up, 1-year post intervention follow-up
  Self-report measure of positive and negative affect (scale 1-6 with higher scores indicating higher affect levels)
Change in School Engagement and Belonging | baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline), 6-month post intervention follow-up, 1-year post intervention follow-up
  Self-report measure of engagement with schoolwork and belonging in school (scale 1-5 with higher scores indicating higher levels of engagement and belonging)
Change in School Grades and Attendance | baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline), 6-month post intervention follow-up, 1-year post intervention follow-up
  Self-report measure of grades and attendance
Change in Physical Health Questionnaire | baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline), 6-month post intervention follow-up, 1-year post intervention follow-up
  Self-report measure of health outcomes such as sleep and physical symptoms (scale 1-7 with higher scores indicating higher levels of health symptoms)
Change in Humanitarian Egalitarian Scale | baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline), 6-month post intervention follow-up, 1-year post intervention follow-up
  Self-report measure of agreement with humanitarian and egalitarian values (scale 1-5 with higher scores indicating higher levels of agreement)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Boulder, Boulder, Colorado, United States